CLINICAL TRIAL: NCT03383315
Title: Role of Prophylactic Metoclopramide With Tramadol in Trauma Patients: A Randomised, Double Blind Placebo Controlled Trial
Brief Title: Role of Prophylactic Metoclopramide With Tramadol in Trauma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Choo Kim Hoon, Doctor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NMRR-16-1688-32638
Record Dates: First submitted 2017-12-18; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Trauma; Opioid Analgesic Adverse Reaction
MeSH Terms: conditions — Wounds and Injuries | interventions — Tramadol; Metoclopramide

STUDY DESIGN:
Intervention Model Description: Patients are randomized into two groups. One group receives tramadol and metoclopramide, while another group receives tramadol and placebo (normal saline).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study drugs were prepared under sterile conditions by a pharmacist independent to the study and kept in packs.The patients recruited were randomized to receive one of the study packs. The study pack were numbered by the pharmacist, who used a computer-generated random number sequence to assign treatment allocations. The allocation list was kept by the pharmacist. Treatment allocations were revealed only after study completion, when all outcome measurements had been performed and recorded by the investigator in the study database.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Intravenous tramadol 50mg + intravenous metoclopramide 10mg
  Interventions: Drug: Tramadol; Drug: Metoclopramide
- Group 2 (Active Comparator): Intravenous tramadol 50mg + placebo (normal saline)
  Interventions: Drug: Tramadol; Drug: Placebo

INTERVENTIONS:
Drug: Tramadol — One dose of intravenous tramadol 50mg
Drug: Metoclopramide — One dose of intravenous metoclopramide 10mg
  Arms: Group 1
Drug: Placebo — Sodium chloride 0.9%
  Arms: Group 2

SUMMARY:
Tramadol is widely used as analgesic in trauma patients. However, it causes side effects, most notably nausea and vomiting. This study aim to determine the role of prophylactic metoclopramide in preventing tramadol induced nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older on day of presentation to ETD SGH
* Sustained from traumatic injuries of extremities (Fracture of hand & wrist, radius, ulna, humerus, femur, tibia, fibula and/or foot & ankle; laceration wounds of extremities; soft tissue injury)
* Patient who is able to give consent

Exclusion Criteria:

* Known allergy to metoclopramide
* Concurrently taking medication with anti-emetic effect, including antihistamines, phenothiazines and dopamine antagonists.
* A history of vomiting since time of injury
* Patients who had already received tramadol or metoclopramide in the previous 8 hours prior to arrival at ETD
* Below age of 18 on day of presentation, or patients who could not consent to the study
* Any alteration in level of consciousness
* Hemodynamic instability or primary diagnosis requiring time critical intervention
* Pregnancy or lactation
* History or known case of vertiginous disorder
* Currently undergoing chemotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Nausea severity scale | One hour
  Change in rating of nausea severity on Visual Analogue Scale 60 minutes after administration of the study drugs. VAS is a standard 100mm line marked "no nausea" at the left end and "worst nausea imaginable" at the right end. Minimum clinically significant difference is defined for this study as 20 mm increment.

SECONDARY OUTCOMES:
Vomiting | One hour
  Number of episodes of vomiting 60 minutes after administration of study drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Sarawak General Hospital, Kuching, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No